CLINICAL TRIAL: NCT01690507
Title: Phase 1/2 Study of Decitabine Combined With Modified CAG Followed by HLA Haploidentical T Cell Infusion in Treating Elderly Patients With Intermediate-high Risk Myelodysplastic Syndrome(MDS) or Acute Myeloid Leukemia(AML）
Brief Title: Decitabine Combining Modified CAG Followed by HLA Haploidentical Peripheral Blood Mononuclear Cells Infusion for Elderly Patients With Acute Myeloid Leukemia(AML）
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Chinese PLA General Hospital (Other)
Collaborators: Navy General Hospital, Beijing (Other)
Responsible Party: Principal Investigator, Li Yu, Director of Department of Hematology and BMT Center, Chinese PLA General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CN301-XYK-001
Record Dates: First submitted 2012-09-19; First posted 2012-09-21 (Estimated); Last update posted 2016-02-25 (Estimated); Status verified 2016-02

CONDITIONS: MDS; AML
Keywords: demethylating agent; immunogenicity
MeSH Terms: interventions — Decitabine; Cytarabine; aclacinomycins; Granulocyte Colony-Stimulating Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- DCAG plus HLI (Other)
  Interventions: Drug: Decitabine; Drug: Cytarabine; Drug: aclacinomycin; Drug: Granulocyte colony-stimulating factor; Other: HLA haploidentical mononuclear cells infusion

INTERVENTIONS:
Drug: Decitabine — 20 mg/m²/day for 5 days
Drug: Cytarabine
Drug: aclacinomycin
Drug: Granulocyte colony-stimulating factor
  Other Names: G-CSF
Other: HLA haploidentical mononuclear cells infusion
  Other Names: DLI

SUMMARY:
Demethylating agent decitabine enhances the immunogenicity of leukemia cells by inducing the expression of cancer testis antigens (CTAs),MHC class I and II molecules,costimulatory molecules and adhesion molecules. The leukemias cells treated by decitabine will become more sensitive to the following adoptive T cell therapy.

ELIGIBILITY:
PATIENT Inclusion Criteria:

* Must have a diagnosis of MDS-RAEB or AML based on 2008 World Health Organization (WHO) classification of myeloid malignancies
* Must have life expectancy >= 3 months
* Must have the ability to observe the efficacy and events
* Must have no accompany therapy(including steroid)
* Patient must have ability to understand and willingness to provide written informed consent prior to participation in the study and any related procedures being performed
* Must have an Eastern Cooperative Oncology Group (ECOG) performance status =< 3
* Must have haploidentical donor

DONOR Inclusion Criteria:

* Must have signed the standard informed consent form; if sufficient cryopreserved cells remain from a previous donation, no additional donation or consent is required
* Both men and women and members of all races and ethnic groups are eligible for this trial

PATIENT Exclusion Criteria:

* Must not have an advanced malignant hepatic tumor
* Must not receive any other forms of chemotherapy after cell infusion during the treatment protocol
* Must not be receiving any other investigational agents within 14 days of first dose of study drug
* Must not have uncontrolled intercurrent illness including ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, or psychiatric illness/social situations that would limit compliance with study requirements
* Must not be pregnant or breastfeeding; pregnant women are excluded from this study because decitabine is a Category D agent with the potential for teratogenic or abortifacient effects; because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with decitabine, breastfeeding should be discontinued if the mother is treated with decitabine; these potential risks may also apply to other agents used in this study
* Must not have a history of allergic reactions attributed to compounds of similar chemical or biologic composition to decitabine or other agents used in the study
* Must not have a known or suspected hypersensitivity to decitabine
* Must not be human immunodeficiency virus (HIV)-positive and on combination antiretroviral therapy; these patients are ineligible because of the potential for pharmacokinetic interactions with decitabine; in addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy; appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated

DONOR Exclusion Criteria:

* Must not have any underlying conditions which would contra-indicate apheresis
* Must not be pregnant

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2012-11; Primary Completion 2015-05 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
CR rate | 3 months

SECONDARY OUTCOMES:
overall survival | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Li Yu, M.D. Ph.D., Principal Investigator — Chinese PLA General Hospital
Locations (2):
- China (2):
  - Navy General Hospital, Beijing, Beijing Municipality
  - Chinese PLA General Hospital, Beijing

REFERENCES:
- [Derived] Jing Y, Jin X, Wang L, Dou L, Wang Q, Yao Y, Lian S, Zhou J, Zhu H, Yao Z, Gao L, Wang L, Li Y, Bai X, Fang M, Yu L. Decitabine-based chemotherapy followed by haploidentical lymphocyte infusion improves the effectiveness in elderly patients with acute myeloid leukemia. Oncotarget. 2016 Aug 10;8(32):53654-53663. doi: 10.18632/oncotarget.11183. eCollection 2017 Aug 8. PMID 28881839